CLINICAL TRIAL: NCT01293123
Title: Raltegravir Cerebrospinal Fluid Pharmacodynamic Study in HIV-Infected Individuals
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Did not meet enrollment goals
Sponsor: University of California, San Diego (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Scott Letendre, Associate Professor of Medicine, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-0067
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Results first posted 2019-10-31 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: HIV
Keywords: HIV; raltegravir; cerebrospinal fluid
MeSH Terms: interventions — Raltegravir Potassium; Tenofovir; Emtricitabine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raltegravir (Experimental)
  Interventions: Drug: Raltegravir
- Efavirenz (Active Comparator)
  Interventions: Drug: Efavirenz

INTERVENTIONS:
Drug: Raltegravir — raltegravir 400 mg PO twice daily
  Other Names: tenofovir disoproxil fumarate 300 mg PO once daily; emtricitabine 200 mg PO once daily
  Arms: Raltegravir
Drug: Efavirenz — efavirenz 600 mg PO once daily
  Other Names: tenofovir disoproxil fumarate 300 mg PO once daily; emtricitabine 200 mg PO once daily
  Arms: Efavirenz

SUMMARY:
The primary aim of this study is to determine the effects of the HIV integrase inhibitor, raltegravir, in cerebrospinal fluid (CSF). This will be accomplished by collecting CSF before and after initiation of either raltegravir or another antiretroviral, efavirenz, each in combination with two other antiretrovirals. Assessments will include HIV RNA levels (viral load), neuropsychological testing, mood assessments, and quality of life assessments.

DETAILED DESCRIPTION:
Cognitive disorders continue to be a common complication of HIV disease even though potent antiretroviral drugs can reduce HIV below detectable levels and restore immune function. Concentrations of most antiretrovirals in the nervous system are only a fraction of concentrations in blood. As a result, HIV can continue to be present in the nervous system when it is below detection in blood. A recently approved drug, raltegravir, reaches therapeutic concentrations in cerebrospinal fluid and may be effective at controlling HIV replication in the primary target cells in the brain, macrophages and microglia. Based on this, raltegravir may be a particularly effective drug for treating HIV disease in the nervous system. The purpose of this study is to determine the effects of raltegravir in the nervous system by measuring HIV in the CSF (via lumbar puncture, also known as spinal taps) before and after initiation of raltegravir-containing antiretroviral therapy. CSF is an accessible fluid that provides a window into brain processes, including HIV replication and inflammation. The potency of raltegravir will be estimated by calculating the change in HIV viral load in CSF over time. These changes will be compared to those following initiation an efavirenz-containing regimen in a separate group of individuals. Two additional drugs (tenofovir disoproxil fumarate, emtricitabine) will be combined with either raltegravir or efavirenz. Neuropsychological performance, mood, sleep and quality of life assessment will also be compared. Participants will be randomly assigned to either raltegravir- or efavirenz-containing therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18-65 years;
2. Integrase inhibitor-naive subjects with clinical indication to initiate RAL under the supervision of their HIV care provider;
3. Baseline detectable HIV-1 RNA levels ≥ 5000 copies/mL in plasma and ≥ 500 copies/mL in CSF;
4. Absolute T-cell CD4+ subset between 200-500/mm3
5. Individual willing to undergo serial lumbar punctures as outlined in study evaluations;
6. Subject able to give informed consent to all study procedures (if cognitively impaired, the individual must pass an evaluation to ensure adequate comprehension of the consent document and procedures);
7. Susceptibility to all study drugs on Monogram Biosciences PhenoSense GT assay.

Exclusion Criteria:

1. Contraindication to lumbar puncture, such as current coagulopathy, thrombocytopenia (platelets below 50,000/µL), or use of anticoagulants;
2. Cognitive, psychiatric, or substance use disorders or any other medical conditions that would interfere with study participation, in the opinion of the investigator;
3. Major opportunistic infections (e.g., pneumonia, tuberculosis) within 30 days;
4. Use of prescribed drugs with known substantial interactions with the study drugs;
5. Positive HCV serology;
6. HIV-associated dementia/Global Deterioration Scale ≥4;
7. Pregnancy;
8. Serum creatinine higher than 2.0 mg/dL;
9. Total bilirubin or alanine or aspartate transaminases more than 3 times the upper limit of normal

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2011-12; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Letendre, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Antiviral Research Center, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Raltegravir | Efavirenz
Started | 1 | 1
Completed | 1 | 0
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raltegravir | Efavirenz | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (0) | 36 (0) | 31 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Cerebrospinal Fluid HIV RNA Levels
Description: Slope of decline of HIV RNA levels in CSF over time
Time Frame: 180 days
Population: Insufficient enrollment for data analysis
Arm/Group | Raltegravir | Efavirenz
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Neuropsychological Performance
Description: Change in neuropsychological performance over 180 days
Time Frame: 180 days
Population: Insufficient enrollment for data analysis
Arm/Group | Raltegravir | Efavirenz
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Measure of Mood
Description: Change in mood over 180 days
Time Frame: 180 days
Population: Insufficient enrollment for data analysis
Arm/Group | Raltegravir | Efavirenz
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Measure of Sleep
Description: Change in self-reported sleep performance over 180 days.
Time Frame: 180 days
Population: Insufficient enrollment for data analysis
Arm/Group | Raltegravir | Efavirenz
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Measure of Quality of Life
Description: Change in self-report quality of life over 180 days
Time Frame: 180 days
Population: Insufficient enrollment for data analysis
Arm/Group | Raltegravir | Efavirenz
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Raltegravir | Efavirenz
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1

LIMITATIONS AND CAVEATS:
Insufficient enrollment for data analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes